CLINICAL TRIAL: NCT00865813
Title: Biopsy Incisional With Trepan in Periocular Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Suzana Matayoshi, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1143/07
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Tumor
Keywords: Punch biopsy,; periocular; tumors.
MeSH Terms: conditions — Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Punch Biopsy (Experimental)
  Interventions: Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Punch Biopsy — 1. Instillation of anesthetic eye drops.
  2. Asepsis
  3. Placement of surgical cloths and drapes
  4. Infiltration of the involved region with anesthetic solution plus adrenalin in1:200.00 dilution.
  5. Trephination of the most typical area of the lesion with a punch (2mm in diameter) of stainless steel by applying gentle pressure and twisting the trephine until its introduction into the suspicious lesions
  6. Removal of the excised tissue with the aid of an insulin needle or conjuntival forceps, the base then bein cut with an number 11 surgical blade
  Other Names: Punch 2 mm; Biopsy

SUMMARY:
The purpose of this study was to identify accuracy rates of 2mm punch biopsy technique in diagnosing periocular malignancy.

DETAILED DESCRIPTION:
In each case, the histology obtained at biopsy was compared with that identified at the time of tumor excision.

ELIGIBILITY:
Inclusion Criteria:

* All lesions were initially examined at the slitlamp, after which lesions with malignant characteristics such as texture, size or color alterations asociated with ulceration, prominent borders or elevated contours, irregular borders, telangiectasias or loss of eyelashes were included.

Exclusion Criteria:

* Lesions with not malignant characteristics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
accuracy, positive predictive value, negative predictive value, sensitivity, specificity | In each case, the histology obtained at biopsy was compared with that identified at the time of tumor excision.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel C Carneiro, Principal Investigator — University of Sao Paulo - Hospital das Clinicas